CLINICAL TRIAL: NCT02515136
Title: Stimulus-response Associations in Parkinson's Disease Patients
Brief Title: Stimulus-response and Parkinson's Disease (SRlearning)
Acronym: SRlearning
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: JBL_2014-29
Record Dates: First submitted 2015-07-30; First posted 2015-08-04 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parkinson's disease (Experimental): Parkinson's disease patients
  Interventions: Behavioral: Stimulus-response
- Controls (Other): Healthy volunteers paired with Parkinson's disease patients on sex and age group, whose data will be extracted from a CNRS existing database
  Interventions: Behavioral: Stimulus-response

INTERVENTIONS:
Behavioral: Stimulus-response — See summary

SUMMARY:
In a computerized experiment, visual stimuli will be presented to the parkinson's disease patients and to the controls. They will respond to each image by acting on the keyboard in a specific manner. Each participant will repeat that task 384 times per session. A break will be inserted every 12 tests so that participants can rest.

The experiment consists of three sessions. Each image will be presented three times. For the first two presentations it is assumed that a link will be created between the image and the task, and the image and action. In the third presentation, the same task and the same action will be maintained or will be swapped. In this way, It can be checked whether associations thus generated will affect the performance of the participants when tasks and actions will be incongruent.

ELIGIBILITY:
Inclusion Criteria:

* Patient : Parkinson's disease Controls: healthy volunteers paired to patients on sex and age group

Exclusion Criteria:

* Other neurological condition
* Known pregnancy or breastfeeding woman
* No medical insurance coverage
* Person under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Reaction time (second) | immediate

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France